CLINICAL TRIAL: NCT03854084
Title: Effect of the Cranial Osteopathic Techniques on the Symptoms of Benign Paroxysmal Positional Vertigo
Brief Title: Cranial Osteopathic Techniques on the Symptoms of Benign Paroxysmal Positional Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laiana Sepúlveda de Andrade Mesquita (Other)
Responsible Party: Sponsor-Investigator, Laiana Sepúlveda de Andrade Mesquita, Senior Researcher, Universidade Estadual do PiauÍ
Organization: Universidade Estadual do PiauÍ (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDAAA 801
Record Dates: First submitted 2019-02-17; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The cranial osteopathic techniques
  Interventions: Other: The cranial osteopathic techniques
- control group (Sham Comparator): Control group
  Interventions: Other: Control group

INTERVENTIONS:
Other: The cranial osteopathic techniques — Technique of the temporal bones in favor of the free movement. Ear Pull technique: the hands of the osteopath holds the auricle of the individual with the thumb, index and the middle finger in a tweezer shape and with the elbows resting over the stretcher. Ruddy technique: The osteopath puts the thumbs on the eyelid of each eyeball.
  Arms: Intervention group
Other: Control group — Simulation of the techniques was used in the interventional group
  Arms: control group

SUMMARY:
The benign paroxysmal positional vertigo (BPPV) is a type of peripheral vertigo characterized by the accumulation of otoliths debris, which are particles resulted from the condensation of endolymph in the inner ducts of semicircular canals (duct lithiasis or canalithiasis). In order to detect the BPPV, a simple test is utilized. The Dix-Hallpike test consists in lay the individual in a quick change in the position of the head. The maneuver is performed, essentially, towards the side in which the patient alleges dizziness in the course of the change in the position of the head. If the individual report vertigo related or no to nystagmus, the test is considered as positive . The osteopathy is a science, which has specific methods of diagnosis and treatment, and has begun to be developed by the physician Andrew Taylor Still at the end of 19th century, which aim is to rebalance the activities of the organism. Accord to the osteopathy science, all the physiological structures in the organism integrating and requires functional and structural harmonization in order to improve the health of the whole body. The main objective of the treatment is to obtain the intertissue mobility, which is considered by osteopathy as a somatic dysfunction, when it is restricted. Samutt confirms that cranial dysfunction of the temporal bones in internal/external rotation may modify the orientation of the semicircular canals, provoking vertigo. Liem propose that the mobilization of the eyeball may be a sensory stimulus of the vestibulo-ocular pathways. For him, maneuvers to the eyeball assists to balance the tonus of extraocular muscles and creates fascial influences on the optic nerve and the oculomotor, and, thus, stimulates the vestibular nuclei. It also suggests that the tension of the cerebellar tentorium and the mobilization of the temporal bones have effects on the structures that composes the vestibule. Thereby, the present work investigated the effect of the cranial osteopathic techniques on the Benign Paroxysmal Positional Vertigo.

DETAILED DESCRIPTION:
The vertigo is the illusive sensation of motion around the ambiance, results in disorders in the physical and social health of the patient due to difficulty in movement and coordination (CAMPOS et al, 2003) and it is classified as one of the four types of dizziness: syncope, disequilibrium, non-specific dizziness or lightheadedness and vertigo. The vertigo may have peripheral and central causes . In peripheral vertigo, its source situated in the labyrinth or in vestibular nerve, until your entrance in vestibular nuclei. In the central vertigo, its origin located in the vestibular nuclei, in brainstem or cerebellum.

Vestibular, visual and proprioceptive systems provides the balance. The vestibular system finds in the inner ear and consists of bony and membranous labyrinths. The entire set is placed in the petrous part of the temporal bones where it is located the cochlea (structure involved in hearing), three semicircular canals and the vestibule. The bony labyrinth contains the perilymph, which has electrolytic function analogous to extracellular wall, additionally, fulfills the tympanic and vestibular cavities. The membranous labyrinth consists of endolymph and ciliated structures sensitive to its movement (otoliths), located in the ampulla (terminal portion of the semicircular canals) which are susceptible to positional changes in the head . The vestibule has sensory organs (utricle and saccule) which assists the ciliated cells monitoring the position of the head. Such structures contain calcium carbonate crystals, responsive to acceleration and gravity effect.

Pereira highlights that vestibulo-ocular reflex uses the information from the sensory organs of the inner ear - saccule and utricle - to generate compensatory movements to position of the head on extraocular muscles. The anterior inferior cerebellar artery, a branch originate in the basilar artery, supplies the whole vestibular system.

With regards to balance, it is significantly important understand the anatomic relation of the vestibule with the vestibular reflexes which consists the visual and proprioceptive systems. All the information derived from the semicircular canals and from the otoliths (saccule and utricle) reaches the cerebellum and the vestibular nuclei as of afferent fibers of vestibular nerve. The processing and integration of central nervous system with the afferent signals from vestibular, visual and proprioceptive systems allows to produce the vestibulo-ocular (maintains the compensatory movement of the eyes regarding the movement from the head), vestibulospinal (produces dynamic and static strategies related to posture), cervico-ocular (steadies the neck through information received from vestibule) reflexes.

The benign paroxysmal positional vertigo (BPPV) is a type of peripheral vertigo characterized by the accumulation of otoliths debris, which are particles resulted from the condensation of endolymph in the inner ducts of semicircular canals (duct lithiasis or canalithiasis). This process induces an abnormal acceleration of endolymph, providing a response to central nervous system that the head is spinning leading to the symptoms and characteristics of BPPV: sudden changes in the position of the head, such as rolling over the bed or tilting the head may causes quick episodes of vertigo, which lasts between 30 seconds to 2 minutes following, or not, of nystagmus, not associated with auditory problems.

In order to detect the BPPV, a simple test is utilized. The Dix-Hallpike test consists in lay the individual in a quick change in the position of the head. The maneuver is performed, essentially, towards the side in which the patient alleges dizziness in the course of the change in the position of the head. If the individual report vertigo related or no to nystagmus, the test is considered as positive.

The osteopathy is a science, which has specific methods of diagnosis and treatment, and has begun to be developed by the physician Andrew Taylor Still at the end of 19th century, which aim is to rebalance the activities of the organism. Accord to the osteopathy science, all the physiological structures in the organism integrating and requires functional and structural harmonization in order to improve the health of the whole body. The main objective of the treatment is to obtain the intertissue mobility, which is considered by osteopathy as a somatic dysfunction, when it is restricted.

The osteopathy concerning to skull had their first records by William G. Sutherland, and it is treated as an extension of the principles of the applied osteopathy in the cranial bones. In his study of the so-called Craniosacral Therapy, Sutherland presuppose that exists a primary respiratory movement, which depends on rhythmic pressure changes induced by alteration of the venous pressure inside the medullary cavity, which causes the pressure of the cerebrospinal fluid varies, of the tensions in the reciprocal membranes, which are the falx cerebri (sagittal) and the cerebellar tentorium (transverse). These membranes are connected to sacrum through the dura mater.

Samutt confirms that cranial dysfunction of the temporal bones in internal/external rotation may modify the orientation of the semicircular canals, provoking vertigo. Liem propose that the mobilization of the eyeball may be a sensory stimulus of the vestibulo-ocular pathways. For him, maneuvers to the eyeball assists to balance the tonus of extraocular muscles and creates fascial influences on the optic nerve and the oculomotor, and, thus, stimulates the vestibular nuclei. It also suggests that the tension of the cerebellar tentorium and the mobilization of the temporal bones have effects on the structures that composes the vestibule.

Thereby, the present work investigated the effect of the cranial osteopathic techniques on the Benign Paroxysmal Positional Vertigo.

ELIGIBILITY:
Inclusion Criteria:

* Were included in the study male and female individuals with age range between 25 and 45 years, BPPV positives.

Exclusion Criteria:

* The exclusion criteria were being in use of any medication for vertigo treatment and the presence of any infectious pathology or deformity in the inner ear.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Dix-Hallpike test | 5 weeks
  consists in provoke a sudden change of position: with the eyes open and looking forward; shifts quickly from the sitting position with the head leaning 45 degrees to one of the sides, with the head hanging. Sits again and perform the same procedure to the opposite side. The maneuver is executed initially to the side where the patient related dizziness while the change of the position of the head. When the individual is not able to recognize in which side the dizziness occurs, the investigators have begun the maneuver on the right side, in order to standardize the test. All the stages of the test must be performed with 40 seconds gap (CAMPOS et al., 2006; HERDMAN; 2003).

CONTACTS AND LOCATIONS:
Locations (1):
- Laiana Sepúlveda de Andrade Mesquita, Teresina, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: Undecided